CLINICAL TRIAL: NCT00080899
Title: A Phase II Trial of Fenretinide (4-HPR) in Biochemically Recurrent, Hormone Naive Prostate Cancer
Brief Title: Fenretinide in Treating Patients With Biochemically Recurrent Hormone-Naïve Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02833; PHII-47; N01CM62209 (NIH); CDR0000357312 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fenretinide

ARMS (1):
- Treatment (fenretinide) (Experimental): Patients receive oral fenretinide twice daily on days 1-7. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fenretinide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fenretinide — Given orally
  Other Names: fenretinimide; McN-R-1967
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well fenretinide works in treating patients with biochemically (rising PSA level) recurrent hormone-naïve (no previous hormone therapy) prostate cancer. Drugs used in chemotherapy, such as fenretinide, work in different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the PSA response in prostate cancer patients with only biochemical recurrence after local curative therapy who are then treated with fenretinide (4-HPR).

II. To assess PSA doubling time as a measure of disease activity, time to PSA progression in prostate cancer patients receiving fenretinide.

III. To evaluate the qualitative and quantitative toxicities of this agent in this patient population.

IV. To evaluate pharmacokinetic studies on the bioavailability of 4-HPR in this patient population.

OUTLINE: This is a multicenter study. Patients are stratified according to prior therapy (surgery vs radiotherapy and/or brachytherapy vs both), stage at diagnosis (organ confined vs extra-capsular extension vs lymph node positive), Gleason score at diagnosis (2-4 vs 5-6 vs 7-10), and prostate-specific antigen level at diagnosis (0-4 ng/mL vs 4.1-10 ng/mL vs > 10 ng/mL).

Patients receive oral fenretinide twice daily on days 1-7. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically or cytologically confirmed history of adenocarcinoma of the prostate
* Patients must have a rising PSA, following a nadir value of < 4 ng/mL for patients treated with primary radiation and < 0.3 ng/mL for patients treated with radical prostatectomy, with no clinical or radiographic evidence of metastatic disease; the rising PSA must be confirmed by two consecutive increases, separated by at least 2 weeks; the absolute PSA value must be > 2.0 ng/mL, and the increment of increase must be at least 0.5 ng/mL above the nadir
* Following radical prostatectomy, patients can have received adjuvant radiation therapy for positive margins or pT3 disease; patients may also have received radiation therapy for local recurrence, provided that they subsequently have a rising PSA after a new PSA nadir of < 4ng/mL
* Bone scan negative for metastatic disease within 4 weeks prior to registration
* Patients must have a performance status of 0, 1, or 2
* The effects of fenretinide on fetal conception and development at the recommended therapeutic dose are unknown; for this reason, men enrolled in this trial must agree to use adequate contraception prior to study entry and for the duration of study participation
* Peripheral absolute neutrophil count (ANC) >= 1000/μL
* Platelet count >= 100,000/μL (transfusion independent; defined as: without transfusion for 3 weeks prior to obtaining study entry value)
* Hemoglobin >= 8.0 gm/dL (may receive RBC transfusions or exogenous erythropoietin)
* Life expectancy of greater than 3 months
* Serum creatinine =< 1.5 gm/dL
* Creatinine clearance or radioisotope GFR >= 50 ml/min/m2
* Total bilirubin =< 1.5 mg/dL
* SGOT (AST) and SGPT (ALT) < 2.5 x normal
* Patients with seizure disorders may be enrolled if on anticonvulsants and well controlled
* CNS toxicity =< Grade 2
* Patient must be able to consume the entire intact capsule(s) in the dosage prescribed for body surface area
* Triglycerides are less than 300mg/dl
* All patients will have malignancy confirmed by review of their biopsy specimens by the Division of Pathology of the City of Hope National Medical Center, the University of Southern California/LA County/Norris Comprehensive Cancer Center, or the University of California at Davis
* In patients who received radiotherapy, the absolute increase of PSA must be at least 2ng/ml to account for the "bounce" phenomenon

Exclusion Criteria:

* Patients with evidence of metastatic disease
* PSA progression not verified by sequential rising PSA as discussed in Eligibility section
* Inability to take oral fenretinide
* Patients who have had prior cytotoxic chemotherapy or androgen ablative therapy
* Patients with history of receiving, or current administration of, chemotherapeutic agents, biological response modifiers, or corticosteroids; patients are permitted to have received up to 9 months of neoadjuvant or adjuvant hormone ablation in conjunction with their primary definitive therapy; androgen deprivation must have been completed at least one year prior to registration; no complementary or alternative therapy (e.g. St. John's Wort, PC-SPES, or other herbal remedies taken for the purpose of treating prostate cancer) may be given during protocol treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fenretinide (i.e. retinoids)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of any site, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* Patients should not take any drugs suspected of causing pseudotumor cerebri, which include tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, amiodarone, or vitamin A
* Patients may have received one prior investigational anti-cancer agent
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from this study because of possible pharmacokinetic interactions with fenretinide; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients should not concurrently take medications that may potentially act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, or p-glycoprotein (MDR1) or MRP1 drug/lipid transporters, such as: cyclosporine A or analogue; verapamil; tamoxifen or analogue; ketoconazole, chlorpromazine; RU486; indomethacin; or sulfinpyrazone
* Patients with known uncontrolled hypertriglyceridemia resulting in pancreatitis are excluded from study; patients with fasting triglycerides equal to or greater then 300mg/dl should start on medical treatment for hypertriglyceridemia (ex. fibrate derivatives); fenretinide will only be started when triglycerides are less than 300mg/dl
* Patients with known retinopathy from any source are excluded from the protocol as elevated ceramide levels from Fenretinide may exacerbate and/or lead to permanent retinal damage in this population
* Patients taking antioxidant supplements (vitamin C or E) must discontinue use before being eligible for protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Principal Investigator — University of Southern California, Norris
Locations (1):
- University of Southern California, Norris, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients received Fenretinide (N-(4-hydroxyphenyl) retinamide [4-HPR]) at a dose of 900 mg/m2 twice daily for the maximal practical dose of 1800 mg/m2/day for 1 week, every 3 weeks, for 1 year.
Period: Overall Study
Arm/Group | Arm 1
Started | 23
Completed | 22
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 69 [53 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: PSA normalization (PSA-N) was recorded as the best PSA response when a PSA level was undetectable (< 0.1 ng/ml), and was then subsequently confirmed by a second measurement ≥ 4 weeks later. PSA partial response (PSA-PR) was recorded if the PSA decreased by ≥ 50% from pre-treatment or baseline values and was confirmed by a second measurement made ≥ 4 weeks later. Response = PSA-N + PSA-PR.
Time Frame: Baseline to 5 years
Measure: Number; unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 22
participants | 0

2. Secondary Outcome: Time to PSA Progression
Description: Was summarized using the product-limit (Kaplan-Meier) method. In patients whose PSA levels initially decreased, PSA progression was defined as a 25% increase over the nadir (postenrollment PSA value up to that point), and an increase in the absolute value in the PSA value of 5 ng/mL, relative to the lowest postenrollment PSA value up to that point, including the baseline PSA level - and which was confirmed by second value 3-4 weeks later. A best response of PSA-PD was recorded for those patients who did not achieve a confirmed PSA-N or PSA-PR and who experienced PSA progression within 3 months of start of treatment.
Time Frame: From the start of treatment until the date of the first documentation of PSA progression, assessed up to 5 years
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 23
months | 4.6 [3.2 to 8.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 2 years and 9 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 22/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=23)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (23)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Dry eye syndrome (Eye disorders) | 3 (15)
Eye disorder (Eye disorders) | 2 (2)
Flashing vision (Eye disorders) | 8 (51)
Night blindness (Eye disorders) | 10 (45)
Photophobia (Eye disorders) | 5 (13)
Proptosis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (6)
Cheilitis (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 4 (9)
Diarrhea (Gastrointestinal disorders) | 8 (30)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (18)
Nausea (Gastrointestinal disorders) | 5 (11)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 3 (22)
Flu-like symptoms (General disorders) | 1 (1)
Irritability (General disorders) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 3 (11)
Aspartate aminotransferase increased (Investigations) | 3 (11)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (7)
Hyperbilirubinemia (Investigations) | 4 (17)
Hypercholesterolemia (Investigations) | 2 (5)
Lipase increased (Investigations) | 3 (5)
Lymphopenia (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (17)
Anorexia (Metabolism and nutrition disorders) | 2 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 9 (24)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 3 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (16)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (18)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (9)
Headache (Nervous system disorders) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (46)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less